CLINICAL TRIAL: NCT07026656
Title: Pre-clinical Diagnosis Using Integrated Microbial and Host Response Signatures to Improve Outcomes From Ventilator-associated Pneumonia in Critically Ill Children
Acronym: VAP-Dx
Status: Recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nazima Pathan, FRCPCH PhD, University of Cambridge
Other Study IDs: IRAS number: 333103
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: Respiratory Tract Infection; Immunology; Genomics; Paediatric Intensive Care Unit (PICU)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endotracheal Aspirate Oropharyngeal Swab Heparinized Blood PAXgene Whole Blood In Cytodelic Stabilizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ventilator Associated Pneumonia Group: Critically ill children who develop VAP during their PICU journey will be assigned to the VAP group
- Non-Ventilator Associated Pneumonia Group: All patients who fit eligibility criteria for study and do not go on to develop VAP

SUMMARY:
Ventilator-associated pneumonia (VAP), defined as pneumonia occurring 48 hours after initiation of invasive mechanical ventilation, is insidious in onset and severe in consequence. It is a critical issue affecting 10-20% of the 26,000 children admitted to the paediatric intensive care unit (PICU) each year. Infection typically leads to extended PICU stay, prolonged invasive mechanical ventilation, and increased mortality.

Despite its clinical significance, VAP remains poorly defined, as current diagnosis relies on non-specific criteria and the ability to obtain clinically meaningful cultures. VAP, deviates from conventional pneumonia, potentially originating, from tissue damage, changes to immune processes, and migration of gastrointestinal bacteria into the lung; all associated with prolonged mechanical ventilation. These factors, in combination with the clinical instability of PICU patients, mean that clinicians aggressively start antibiotic therapy despite a paucity of evidence to suggest the best regime. As a result, suspected VAP has been shown to account for nearly 40% of antibiotic exposure in the PICU, which has significant implications on anti-microbial resistance (AMR).

To address these challenges, novel diagnostic therapies are needed to optimise the treatment of VAP. These therapies should utilise our current understanding of the pathophysiology of VAP development, specifically, the infiltration of the lung microbiome by gut and oral bacteria during prolonged mechanical ventilation. To achieve this, molecular testing should be promoted allowing for rapid identification of lung pathogens. There is also growing evidence, for the investigation of predictive biomarkers for VAP available in both the blood and lungs, which when integrated into protocols may enhance diagnostic accuracy. These novel techniques may improve clinical outcomes for affected children while addressing the economic impact of prolonged hospital stays and mitigating AMR risks in PICUs.

ELIGIBILITY:
Inclusion Criteria:

* PICU Admission
* Requires 48 Hours Of Mechanical Ventilation

Exclusion Criteria:

* Imminent death or palliative care pathway planned
* Existing tracheostomy at time of admission
* Known immunocompromised patient
* Patient received a full course of systemic antimicrobials in the previous 6 weeks.
* Known or suspected tuberculosis (TB).

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically Ill Children Requiring Mechanical Ventilation For Greater Than 48 Hours
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Characterise temporal shifts in microbial composition and the corresponding host immune response during prolonged mechanical ventilation | 3 years
  Serial metagenomic profiling of the lung microbiome to establish microbial shifts. Concurrently, cytokines collected from blood and endotracheal aspirates will be taken to assess immune changes.
Characterise the AMR burden in VAP and its role in shaping the microbiome during infection. | 3 years
  Utilise metagenomic sequencing to identify AMR genes present on microbes and relate this to VAP development
Develop statistical and/or machine learning models leveraging these signatures independently, or in combination, to identify putative microbial and host biomarkers for early VAP diagnosis | 3 years

SECONDARY OUTCOMES:
Prevalence of VAP | 3 years
  Number of critically ill children requiring mechanical ventilation who develop VAP compared to those who do not
30 day mortality | 3 years
  Mortality status of patients at 30 days
Time To Extubation | 3 years
  Total Time Intubated
Utilisation Of VAP Prevention Bundle | 3 years
Culture Results | 3 years
  Microbiological Results For Each Patient
Days free of antimicrobial therapy in PICU at 7 days | 3 years
  Days free of antimicrobial therapy during the first 7 days of a patients admission to PICU

CONTACTS AND LOCATIONS:
Overall Officials: Nazima Pathan, FRCPCH PhD, Principal Investigator — Department of Paediatrics, University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient data will be collected and stored on REDcap Safe Haven. All data that is shared will be anonymised to ensure it is not identifiable.